CLINICAL TRIAL: NCT05771350
Title: Hemodiafiltration Versus Hemodialysis in Removal of Indoxyl Sulfate in Chronic Hemodialysis Patients
Brief Title: Online Hemodiafiltration Versus Hemodialysis in Removal of Indoxyl Sulfate in Chronic Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed sary gharib, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 301/2016
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hemodialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- online hemodiafiltration (Experimental)
  Interventions: Procedure: online hemodiafiltration
- high flux hemodialysis (Active Comparator)
  Interventions: Procedure: high flux hemodialysis
- low flux hemodialysis (Active Comparator)
  Interventions: Procedure: low flux hemodialysis

INTERVENTIONS:
Procedure: online hemodiafiltration — 20 patients on regular hemodialysis received online hemodiafiltration
  Arms: online hemodiafiltration
Procedure: high flux hemodialysis — 20 patients on regular hemodialysis received high flux hemodialysis
  Arms: high flux hemodialysis
Procedure: low flux hemodialysis — 20 patients on regular hemodialysis received low flux hemodialysis
  Arms: low flux hemodialysis

SUMMARY:
this study aimed to compare the removal of indoxyl sulphate between hemodiafiltration, high flux hemodialysis and low flux hemodialysis

ELIGIBILITY:
Inclusion Criteria:

* maintenance hemodialysis patients aged more than 18 years

Exclusion Criteria:

* active illnesses, hospitalization, malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
dialytic removal of indoxyl sulpahte | one month when all samples were collected
  assessed by the reduction ration of indoxyl sulphate

IPD SHARING:
Plan to Share IPD: Undecided